CLINICAL TRIAL: NCT01150253
Title: Double Blind Randomised Comparison of Two Preparations, One Enriched in Probiotics and One Without Probiotics (Placebo) in Grass Pollen Allergic Rhinitis Patients, Using a Nasal Provocation Test
Brief Title: Effect of a Probiotic on Grass Pollen Allergic Rhinitis Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Model: Crossover
Other Study IDs: 06.09.NRC
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotic fermented milk (Experimental)
  Interventions: Dietary Supplement: L. paracasei fermented milk
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: L. paracasei fermented milk

INTERVENTIONS:
Dietary Supplement: L. paracasei fermented milk

SUMMARY:
Various studies in animals and humans have shown a potential beneficial effect of probiotics consumption on allergy. However, few studies exist that document their efficacy for upper airways allergies such as allergic rhinitis. The objective of this study is to investigate the effect of short-term oral administration of a Lactobacillus paracasei on a nasal provocation test (NPT) with grass pollen, performed out of pollen season. Adult volunteers with allergic rhinitis are enrolled in a randomized, double-blind, placebo-controlled study, based on two 4-weeks cross-over periods of product consumption (probiotic-fermented milk versus placebo), separated by a washout period of 6-8 weeks. Objective and subjective clinical parameters of NPT as well as systemic and nasal immunological parameters are compared between the two treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 35 years
* history of allergic rhinitis to grass pollen confirmed by either a positive skin prick test (wheal diameter >3 mm) or specific IgE for grass pollen (>0.35 kU/L) as titrated by UniCAP 100 (Pharmacia Diagnostics, Uppsala, Sweden) and no history of perennial rhinitis
* a nasal reaction threshold of 10'000 standardized quality units (SQs)/ml grass pollen or less at the screening phase

Exclusion Criteria:

* any medical condition that could influence the study (pregnancy, viral or bacterial airway infection, active allergic rhinitis)
* uncontrolled asthma (peak expiratory flow <20% of volunteer's best personal value)
* treatment with antihistamine or antibiotic treatment less than two weeks before enrolment or during the trial

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Dates: Start 2006-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: François Spertini, Prof, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Result] Wassenberg J, Nutten S, Audran R, Barbier N, Aubert V, Moulin J, Mercenier A, Spertini F. Effect of Lactobacillus paracasei ST11 on a nasal provocation test with grass pollen in allergic rhinitis. Clin Exp Allergy. 2011 Apr;41(4):565-73. doi: 10.1111/j.1365-2222.2011.03695.x. PMID 21395878